CLINICAL TRIAL: NCT01179477
Title: QuickFlex® μ Model 1258T Left Heart Pacing Lead Post Approval Study
Brief Title: QuickFlex Micro Left Ventricular Lead Post Approval Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD561
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Left heart pacing lead; Cardiac resynchronization therapy (CRT); Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantation of a QuickFlex® μ Model 1258T LV Lead — Implantation of a QuickFlex® μ Model 1258T LV Pacing Lead
  Other Names: LV pacing lead

SUMMARY:
The purpose of this multicenter post-approval study is to evaluate the acute and chronic performance of the QuickFlex® μ 1258T left ventricular (LV) lead.

DETAILED DESCRIPTION:
The primary endpoints of the study are:

* Freedom from LV lead-related complications at 5 years
* LV bipolar capture threshold of St. Jude Medical's QuickFlex®µ 1258T LV Lead measured at 0.5 ms at 5 years

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication per American College of Cardiology/American Heart Association/Heart Rhythm Society guidelines for implantation of a CRT-D system or participated in the QuickFlex® μ1258T (Investigational Device Exemption (IDE) study
* Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate or short term contact with heparin
* Have a life expectancy of less than 5 years due to any condition
* Be less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an approved indication for implantation of a CRT-D system
Sampling Method: Non-Probability Sample
Enrollment: 1930 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay Cohorn, Study Director — Abbott Medical Devices
Locations (77):
- United States (77):
  - Cardiovascular Associates P.C., Birmingham, Alabama
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Heart Center Research, LLC., Huntsville, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - St. Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Northwest Cardiology, Springdale, Arkansas
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Regional Cardiology Associates, Sacramento, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Claudio Bonometti MD, Inc, Santa Barbara, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - Christiana Hospital, Newark, Delaware
  - Shands Jacksonville, Jacksonville, Florida
  - Naushad Shaik, MD, Kissimmee, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Usman R. Siddiqui, MD, Orlando, Florida
  - Orlando Heart Center, Orlando, Florida
  - Brevard Cardiovascular Research Associates, Inc., Rockledge, Florida
  - University of South Florida, Cardiovascular Services, Tampa, Florida
  - Athens Regional Medical Center, Athens, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - The Heart Group, Newburgh, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Mid-America Cardiology Associates, PC, Kansas City, Kansas
  - King's Daughters Medical Center, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Norton Bluegrass Heart Specialists, Louisville, Kentucky
  - Peninsula Cardiology Associates, P.A., Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Trinity Health-Michigan d/b/a Michigan Heart, Ann Arbor, Michigan
  - Thoracic Cardio Healthcare Found. (aka Sparrow Research), Lansing, Michigan
  - MidMichigan Physicians Group, Midland, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Heart Consultants P.C., Omaha, Nebraska
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - Lenox Hill Hospital, New York, New York
  - LeBauer HeartCare, Greensboro, North Carolina
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - Primed Cardiology/Kettering Medical Center Network, Kettering, Ohio
  - Regional Cardiovascular Medical Center, Steubenville, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Toledo Clinic, Toledo, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Tri-State Medical Group Cardiology, Beaver, Pennsylvania
  - Capital Cardiovascular Associates, Camp Hill, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cardiology Consultants, Johnson City, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - The Stern Cardiovascular Foundation, Memphis, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - HeartPlace, Bedford, Texas
  - Advanced Heart Care, Plano, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - McKay-Dee Heart Services, Ogden, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Cardiovascular Associates Ltd, Chesapeake, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
  - St. Mary's Hospital, Madison, Wisconsin
  - Cardiac Rhythm Specialists, S.C., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per the clinical investigation protocol, IDE subjects (n=54) who did not consent to roll over into the post approval study (PAS) at sites participating in the post approval study, were included in primary endpoint analyses. Since these subjects are not enrolled into the PAS, they are not reflected in the participant flow.
Groups:
- Subjects Implanted With a New QuickFlex μ Lead: Subjects implanted with a new QuickFlex μ lead and subjects previously enrolled in the QuickFlex μ IDE study were enrolled into the post-approval study. All successfully enrolled subjects were followed every six months for a period of five years.
Period: Overall Study
Arm/Group | Subjects Implanted With a New QuickFlex μ Lead
Started | 1930
Completed | 843
Not Completed | 1087
Not completed — Death | 542
Not completed — Unsuccessful implant | 80
Not completed — Non-death withdrawal | 438
Not completed — Did not complete final visit | 27

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Implanted With a New QuickFlex μ Lead
Number analyzed (Participants) | 1930
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 529
  Male | 1401
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  American Indian or Alaska Native | 2
  Black or African American | 197
  Hispanic or Latino | 67
  Native Hawaiian/Pacific Islander | 2
  Other | 8
  White | 1646
Region of Enrollment [Number; unit: participants]
  United States | 1930
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percent of blood ejected] — LVEF is percent of blood ejected from left ventricle
  Percent of blood ejected | 25.1 (7.6)
Intrinsic QRS duration [Mean (Standard Deviation); unit: ms] | 152.0 (25.2)
New York Heart Association (NYHA) Classification at Baseline [Count of Participants; unit: Participants] — NYHA Functional Classification has 4 categories:
  Class I (least severe) - no limitation of physical activity Class II - slight limitation of physical activity Class III - marked limitation of physical activity Class IV (most severe) - unable to carry on any phyiscal activity without discomfort
  Participants
    Class I | 19
    Class II | 175
    Class III | 1672
    Class IV | 61
    Unknown | 3
Cardiomyopathy [Count of Participants; unit: Participants]
  Ischemic | 1131
  Non-ischemic | 799

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Alive and Without a Left Ventricular Lead-related Complication
Description: Percent of Participants Alive and Without a Left Ventricular Lead-related Complication at 5 years of follow-up. Per FDA, data from IDE subjects who did not consent to rollover into the post approval study at sites participating in the post approval study, were included in this analysis (see clinical investigational protocol).
Time Frame: 5 years
Population: The analysis population for Primary Endpoint #1 includes newly enrolled and IDE rollover subjects with an attempted implant of the QuickFlex μ LV lead (n=1,930) and subjects from the IDE sites that agreed to participate in the post-approval study, but did not consent to rollover into the post-approval study (n=54), for a total of 1,984 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Implanted With a New QuickFlex μ Lead: Subjects implanted with a new QuickFlex μ lead and subjects previously enrolled in the QuickFlex μ Investigational Device Exemption (IDE) study were enrolled into the PAS study. All successfully enrolled subjects were followed every six months for a period of five years.
Arm/Group | Subjects Implanted With a New QuickFlex μ Lead
Number analyzed (Participants) | 1984
Participants | 1902

2. Primary Outcome: Left Ventricular Bipolar Pacing Capture Threshold
Description: Mean left ventricular bipolar pacing capture threshold measured at 0.5 ms pulse width at 5 years of follow-up
Time Frame: 5 years
Population: Subjects included in this analysis are only those who have left ventricular bipolar pacing capture threshold values reported a the 5-year visit. Of the 843 who completed the 5 year visit, only 774 had analzable data.
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Subjects Implanted With a New QuickFlex μ Lead
Number analyzed (Participants) | 774
Volts | 2.04 (1.6)

ADVERSE EVENTS:
Time Frame: Complications and observations post implant through 5 years
Description: Complications are considered serious adverse events. A complication is an event caused by or associated with the study device, system component(s) and/or procedure that requires invasive intervention (e.g. post-implant lead dislodgement requiring repositioning).
  An observation is an event caused by or associated with the study device, system component(s) and/or procedure that does not require invasive intervention (e.g. over-sensing or loss of pacing capture requiring reprogramming)
Arm/Group | Subjects Implanted With a New QuickFlex μ Lead
All-Cause Mortality (participants affected / at risk) | 542/1930
Serious Adverse Events (participants affected / at risk) | 258/1930
Other Adverse Events (participants affected / at risk) | 512/1930
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted With a New QuickFlex μ Lead (N=1930)
Lead Dislodgement or Migration (Injury, poisoning and procedural complications) | 62 (63)
Diaphragmatic/Phrenic Nerve Stimulation (Injury, poisoning and procedural complications) | 16 (16)
Loss of Capture (Product Issues) | 9 (9)
Elevated Pacing Thresholds (Product Issues) | 8 (8)
Abnormal LV Lead Pacing Impedance <= 200 OHMS or >= 2000 OHMS (Product Issues) | 3 (3)
Dizziness (Injury, poisoning and procedural complications) | 1 (1)
Endocarditis (Injury, poisoning and procedural complications) | 1 (1)
Induced Atrial or Ventricular Arrhythmias (Injury, poisoning and procedural complications) | 1 (1)
Lead Fracture (Product Issues) | 1 (1)
Lead Insulation Damage (Product Issues) | 1 (1)
Pain/Discomfort At Incision Site (Injury, poisoning and procedural complications) | 2 (2)
Premature Battery Depletion (Product Issues) | 8 (8)
Infection (Infections and infestations) | 24 (24) — Procedure Related
Suspected Generator Malfunction (Product Issues) | 4 (4)
Erosion (Infections and infestations) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1)
LV Lead Loss of Capture (Product Issues) | 1 (1)
Twiddler Syndrome (Psychiatric disorders) | 3 (4)
Pericardial Effusion (Injury, poisoning and procedural complications) | 2 (2)
RA Lead Dislodgement or Migration (Product Issues) | 20 (22)
RA Abnormal Lead Impedance (Product Issues) | 4 (4)
RA Lead Insulation Damage (Product Issues) | 4 (4)
RA Loss of Capture (Product Issues) | 2 (2)
RA Atrial Lead Noise (Product Issues) | 1 (1)
RA Cardiac/Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 1 (1)
RA Diaphragmatic/Phrenic Nerve Stimulation (Injury, poisoning and procedural complications) | 1 (1)
RA Elevated Pacing Thresholds (Product Issues) | 1 (1)
RA Oversensing (Product Issues) | 1 (1)
RA Undersensing (Product Issues) | 1 (1)
RV Lead Dislodgement or Migration (Injury, poisoning and procedural complications) | 31 (32)
RV Elevated Pacing Thresholds (Product Issues) | 9 (9)
RV Lead Fracture (Product Issues) | 7 (7)
RV Lead Insulation Damage (Product Issues) | 5 (5)
RV Abnormal Lead Impedance (Product Issues) | 4 (4)
RV Cardiac/Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 3 (3)
RV Loss of Capture (Product Issues) | 2 (2)
RV Cardiac Tamponade (Injury, poisoning and procedural complications) | 1 (1)
RV Endocarditis (Infections and infestations) | 1 (1)
RV Inappropriate Shock (Product Issues) | 1 (1)
RV Infection (Infections and infestations) | 1 (1)
RV Oversensing (Product Issues) | 1 (1)
RV Pectoral Stimulation (Injury, poisoning and procedural complications) | 1 (1)
RV Lead Unable to Defibrillate (Product Issues) | 1 (1)
RV Undersensing (Product Issues) | 1 (1)
Procedure Hematoma/Seroma (Injury, poisoning and procedural complications) | 9 (9)
Procedure Pneumothorax/Hemothorax (Injury, poisoning and procedural complications) | 7 (7)
Procedural Pericardial Effusion (Injury, poisoning and procedural complications) | 3 (3)
Procedural Cardiac/Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 2 (2)
Procedural Cardiac Arrest (Injury, poisoning and procedural complications) | 1 (1)
Procedural Cardiac Tamponade (Injury, poisoning and procedural complications) | 1 (1)
Procedural Deep Vein Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Procedural Device Migration (Injury, poisoning and procedural complications) | 1 (1)
Procedural Guidewire Stuck In LV Lead (Injury, poisoning and procedural complications) | 1 (1)
Procedural Lead Dislodgement or Migration (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pleural Effusion (Injury, poisoning and procedural complications) | 1 (1)
Procedural Skin Injury At PG Pocket (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted With a New QuickFlex μ Lead (N=1930)
LV Lead Elevated Pacing Thresholds (Product Issues) | 214 (221) — LV Lead Related Observations
LV Diaphragmatic/Phrenic Nerve Stimulation (Injury, poisoning and procedural complications) | 145 (164) — LV Lead Related Observations
LV Loss of Capture (Product Issues) | 19 (20) — Lead Related Observations
Abnormal LV Lead Pacing Impedance <= 200 Ω or >= 2000 Ω (Product Issues) | 16 (17) — LV Lead Related Observations
LV Induced Atrial or Ventricular Arrhythmias (Injury, poisoning and procedural complications) | 2 (2) — LV Lead Related Observations
LV Lead Dislodgement or Migration (Injury, poisoning and procedural complications) | 2 (2) — LV Lead Related Observations
LV Cardiac/Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 1 (1) — LV Lead Related Observations
LV Coronary Sinus or Cardiac Vein Thrombosis (Injury, poisoning and procedural complications) | 1 (1) — LV Lead Related Observations
LV Lead Insulation Damage (Product Issues) | 1 (1) — LV Lead Related Observations
System/Pulse Generator Related Therapy For Non-Ventricular Rhythm (Cardiac disorders) | 23 (27) — (System / PG / Other Leads/ Procedure)
System/Pulse Generator Related Failed ICD Shock (Product Issues) | 1 (1) — System / PG / Other Leads/ Procedure
System/Pulse Generator Related Idioventricular Rhythm Preventing Biventricular Pacing (Cardiac disorders) | 1 (1) — System / PG / Other Leads/ Procedure
System/Pulse Generator Related Pacemaker Mediated Tachycardia (Product Issues) | 1 (1) — System / PG / Other Leads/ Procedure
RA Lead Related Oversensing (Product Issues) | 9 (9)
RA Lead Related Abnormal Lead Impedance (Product Issues) | 5 (5)
RA Lead Related Atrial Lead Noise (Product Issues) | 3 (3)
RA Lead Related Elevated Pacing Thresholds (Product Issues) | 3 (3)
RA Lead Related Lead Insulation Damage (Product Issues) | 3 (3)
RA Lead Related Loss of Capture (Product Issues) | 2 (2)
RA Lead Related Lead Dislodgement or Migration (Injury, poisoning and procedural complications) | 1 (1)
RA Lead Related Lead Fracture (Product Issues) | 1 (1)
RA Lead Related Myopotential Sensing (Injury, poisoning and procedural complications) | 1 (1)
RA Lead Related Undersensing (Product Issues) | 1 (1)
RV Lead Related Therapy For Non-Ventricular Rhythm (Cardiac disorders) | 6 (6)
RV Lead Related Abnormal Lead Impedance (Product Issues) | 3 (3)
RV Lead Related Lead Insulation Damage (Product Issues) | 2 (2)
RV Lead Related Bilateral Pleural Effusion (Injury, poisoning and procedural complications) | 1 (1)
RV Lead Related Elevated Pacing Thresholds (Product Issues) | 1 (1)
RV Lead Related Lead Externalization (Product Issues) | 1 (1)
RV Lead Related Myopotential Sensing (Injury, poisoning and procedural complications) | 1 (1)
RV Lead Related Oversensing (Product Issues) | 1 (1)
RV Lead Related Pectoral Stimulation (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Hematoma/Seroma (Injury, poisoning and procedural complications) | 33 (33)
Procedure Related Cardiac/Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 12 (12)
Procedure Related Infection (Infections and infestations) | 4 (4)
Procedure Related Atrial Arrhythmia (Injury, poisoning and procedural complications) | 3 (3)
Procedure Related Pericardial Effusion (Injury, poisoning and procedural complications) | 3 (3)
Procedure Related Bleeding And/or Hemoptysis (Injury, poisoning and procedural complications) | 2 (2)
Procedure Related Cardiac Vein Thrombus (Injury, poisoning and procedural complications) | 2 (2)
Procedure Related Part of The Delivery Tool Was Left In The Coronary Sinus/ Ventricle (Injury, poisoning and procedural complications) | 2 (2)
Procedure Related Pneumothorax/Hemothorax (Injury, poisoning and procedural complications) | 2 (2)
Procedure Related Pulmonary Edema (Injury, poisoning and procedural complications) | 2 (2)
Procedure Related Renal Failure or Injury (Injury, poisoning and procedural complications) | 2 (2)
Procedure Related Acute Left Arm Thrombophlebitis (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Cardiac/Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Decompensated Heart Failure (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Device Incision Erythema (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Excessive Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Frozen Shoulder (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related High DFT's (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Hypotension Requiring Medical Intervention During CRT-D Implant (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Myocardial Infarction (Injury, poisoning and procedural complications) | 1 (1)
Procedure Related Pericarditis (Injury, poisoning and procedural complications) | 1 (1)
Other Therapy For Non-Ventricular Rhythm (Cardiac disorders) | 6 (6)
Other Pericardial Effusion (Injury, poisoning and procedural complications) | 3 (3)
Other Induced Atrial or Ventricular Arrhythmias (Injury, poisoning and procedural complications) | 2 (2)
Other Pulmonary Edema (General disorders) | 2 (2)
Other Infection (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2010-06-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT01179477/Prot_000.pdf